CLINICAL TRIAL: NCT06882694
Title: The Turkish Validity and Reliability of the Kinesthetic Motor Imagery of Pelvic Floor Muscle Contraction Questionnaire
Brief Title: Validity and Reliability of the Kinesthetic Motor Imagery of Pelvic Floor Muscle Contraction Questionnaire in Turkish
Status: Not yet recruiting | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/11-13
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-10

CONDITIONS: Pelvic Floor; Motor İmagery Ability
Keywords: pelvic floor; motor imagery ability; reliability; validity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pelvic Floor Imagery Group
  Interventions: Behavioral: Pelvic Floor Imagery Questionairre

INTERVENTIONS:
Behavioral: Pelvic Floor Imagery Questionairre — This intervention consists of a questionairre

SUMMARY:
The aim of this study is to adapt the questionnaire named "Kinesthetic Motor Imagery of Pelvic Floor Muscle Contraction Questionnaire (KMI-PFQ)" into Turkish in healthy women and to introduce it to the literature as a valid and reliable questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-30 years old
* Understanding and speaking Turkish
* Being willing to participate in the study
* Not having any neurological or orthopedic problems
* Not having any pelvic floor pathology diagnosed by a specialist physician

Exclusion Criteria:

* Having any previous or current pelvic floor pathology
* Not understanding or speaking Turkish

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female participants will be accepted for the study.
Study Population: Female participants between the ages of 18-30 who have no diagnosed pelvic floor dysfunction will be included in the study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10-25 (Estimated); Primary Completion 2025-11-09 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Kinesthetic Motor Imagery of Pelvic Floor Muscle Contraction Questionnaire | 20 minutes
  The KMI-PFQ is a 5-item scale through which women reported their ability and mental effort for imagining pelvic floor muscle contractions.The two dimensions of this instrument (ability and mental effort of the imagined contraction) were scored from zero to 5 for each item. In this imagining ability dimension, responses ranged from zero (the contraction is impossible to feel) to 5 (the imagined contraction is very easy to feel). In the mental effort dimension, the responses ranged from zero (the mental effort to perform the contraction was none to 5 (the mental effort to perform the (imagined) contraction was very intense). Considering that the items for the mental effort dimension are reversed, the maximum score that could be obtained was 25 points for each dimension, with 50 being the maximum possible for the whole questionnaire.

SECONDARY OUTCOMES:
Movement Imagination Questionnaire *MIQ-3 | 20 minutes
  The MIQ-3 developed by Williams et al. will be used to assess individuals' imagery abilities. The HIA-3 is a self-report psychometric measurement method that measures both kinesthetic imagery and visual imagery abilities of individuals. The test consists of 12 items. The test assesses both kinesthetic imagery abilities and visual imagery (internal visual imagery and external visual imagery) abilities of individuals. The test includes 3 different ways of imagining 4 movements. After each imagery action, individuals are asked to rate how easy/difficult it is to perform this mental action. Individuals score their mental actions for Internal Visual Imagery and External Visual Imagery with a 7-point Likert-type scale; 1 = Very hard to see, 7 = Very easy to see; for kinesthetic imagery, 1 = Very hard to feel, 7 = Very easy to feel.
Vividness of Visual Imagery Questionnaire (VVIQ-12) | 10 minutes
  The VVIQ-12 was another instrument we used in validating our KMI-PFQ. The VVIQ is a 12-item self-report scale used to assess the vividness of visual images. The 12 items were structured into four factors: moving space images, familiar images, detailed objects recall, and images creative skill. For each item, the participant can score from 1 to 5 according to how easy it is to generate mental images as clear and realistic as normal vision.

IPD SHARING:
Plan to Share IPD: No